CLINICAL TRIAL: NCT02978885
Title: In Vivo Imaging of Peri-operative (periOP) Destructive Processes in the Lung
Brief Title: Imaging of Peri-operative (periOP) Lung Injury
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Poor enrollment
Sponsor: Columbia University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: AAAR0395; 1R01HL131960-01 (NIH)
Record Dates: First submitted 2016-11-28; First posted 2016-12-01 (Estimated); Results first posted 2021-09-14 (Actual); Last update posted 2021-09-14 (Actual); Status verified 2021-08

CONDITIONS: Acute Lung Injury; Chronic Obstructive Pulmonary Disease (COPD)
Keywords: Acute lung injury; Chronic obstructive pulmonary disease (COPD); Whipple procedures; pancreatico-duodenectomies
MeSH Terms: conditions — Acute Lung Injury; Pulmonary Disease, Chronic Obstructive | interventions — Pancreaticoduodenectomy; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Normal preoperative lung function (Other): Patients with normal lung function undergoing Whipple procedures or other major surgeries will receive an injection of AxV-128 labeled with 99mTc followed by SPECT-CT (AxV-128/Tc SPECT-CT imaging).
  Interventions: Radiation: SPECT-CT imaging; Drug: AxV-128/Tc; Procedure: Whipple procedure; Procedure: Major surgery
- Preoperative COPD (Other): Patients with moderate COPD undergoing Whipple procedures or other major surgeries will receive an injection of AxV-128 labeled with 99mTc followed by SPECT-CT (AxV-128/Tc SPECT-CT imaging).
  Interventions: Radiation: SPECT-CT imaging; Drug: AxV-128/Tc; Procedure: Whipple procedure; Procedure: Major surgery

INTERVENTIONS:
Radiation: SPECT-CT imaging — Injection of AxV-128 labeled with 99mTc followed by SPECT CT
  Other Names: SPECT CT
Drug: AxV-128/Tc — Injection of AxV-128 labeled with 99mTc
  Other Names: 99mTc-rhAnnexin V-128
Procedure: Whipple procedure — A Whipple procedure - also known as a pancreaticoduodenectomy - is a complex operation to remove the head of the pancreas, the first part of the small intestine (duodenum), the gallbladder and the bile duct.
  The Whipple procedure is used to treat tumors and other disorders of the pancreas, intestine and bile duct. It is the most often used surgery to treat pancreatic cancer that's confined to the head of the pancreas. After performing the Whipple procedure, your surgeon reconnects the remaining organs to allow you to digest food normally after surgery. Standard of care.
  Other Names: Pancreaticoduodenectomy
Procedure: Major surgery — Additional surgical procedure(s) that is clinically indicated. Standard of care.
  Other Names: Surgical procedure

SUMMARY:
The aim of study is to determine if 99mTc Annexin V-128 (AxV- 128/Tc) single photon emission computed tomography (SPECT)-computed tomography (CT) can detect perioperative lung injury. The investigators will study patients undergoing major surgery, specifically Whipple procedures (pancreatico-duodenectomies) and compare AxV-128/Tc SPECT-CT scans before and after surgery in Chronic Obstructive Pulmonary Disease (COPD) and non-COPD patients.

DETAILED DESCRIPTION:
Lung injury is commonly not detected unless structural damage has occurred. SPECT-CT scanning using a specific tracer that lights up when it detects apoptosis (programmed cell death) has been used to detect even minor lung injury for example by smoke inhalation in animals and may be more sensitive to detect a less severe injury. The present study aims to study SPECT-CT scan using a tracer for apoptosis, 99mTc Annexin V-128 (AxV- 128/Tc), to detect lung injury after major surgery. Prolonged ventilation during surgery can cause minor lung injury but is usually not clinically detected. The investigators are planning to study 40 patients (20 patients with pre-existing lung disease-COPD and 20 patients with normal preoperative lung function) who are undergoing Whipple operations or other major surgery. The investigators will obtain SPECT-CT scans before and then 2-3 days after surgery and compare the uptake of a radioactive tracer with plasma markers of lung injury (Soluble Receptors for Advanced Glycation End Products (sRAGE), Interleukin 6 (IL-6), Clara-cell 16 and lung surfactant protein D (SP-D) among others). The investigators will ask the subjects to undergo spirometry testing, blood draws and urine collection. In addition, a SPECT-CT scan that lasts approximately 1 hour will be performed prior to surgery and 2-3 days post-operatively (while still hospitalized).

The total effective dose from the combined SPECT and CT scans is 6.2 millisievert (mSv). This effective dose is below what a patient receives during a standard 2 dose rest and stress cardiac nuclear imaging study and well within the range of current clinical nuclear imaging tests. The exact long term risk for development of cancer from diagnostic radiological procedures is currently under debate but all imaging procedures in this study are aimed to keep total radiation burden As Low As Reasonably Achievable (ALARA).

ELIGIBILITY:
Inclusion Criteria:

* Patients with moderate COPD (Global Initiative for Chronic Obstructive Lung Disease (GOLD) stage II: forced expiratory volume 1 (FEV1)/forced vital capacity (FVC) <0.70 and FEV1 50-79% normal) undergoing Whipple procedures or other major surgeries
* Patients with normal lung function undergoing Whipple procedures or other major abdominal surgeries

Exclusion Criteria:

* Age < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2018-06-11 (Actual); Primary Completion 2020-02-05 (Actual); Study Completion 2020-02-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gebhard Wagener, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Normal Preoperative Lung Function: Patients with normal lung function undergoing Whipple procedures or other major surgeries will receive an injection of AxV-128 labeled with 99mTc followed by SPECT-CT (AxV-128/Tc SPECT-CT imaging).
  SPECT-CT imaging: Injection of AxV-128 labeled with 99mTc followed by SPECT CT
  AxV-128/Tc: Injection of AxV-128 labeled with 99mTc
  Whipple procedure: A Whipple procedure - also known as a pancreaticoduodenectomy - is a complex operation to remove the head of the pancreas, the first part of the small intestine (duodenum), the gallbladder and the bile duct.
  The Whipple procedure is used to treat tumors and other disorders of the pancreas, intestine and bile duct. It is the most often used surgery to treat pancreatic cancer that's confined to the head of the pancreas. After performing the Whipple procedure, your surgeon reconnects the remaining organs to allow you to digest food normally after surgery. Standard of care.
  Major surgery: Additional surgical procedure(s) that is clinically indicated. Standard of care.
- Preoperative COPD: Patients with moderate COPD undergoing Whipple procedures or other major surgeries will receive an injection of AxV-128 labeled with 99mTc followed by SPECT-CT (AxV-128/Tc SPECT-CT imaging).
  SPECT-CT imaging: Injection of AxV-128 labeled with 99mTc followed by SPECT CT
  AxV-128/Tc: Injection of AxV-128 labeled with 99mTc
  Whipple procedure: A Whipple procedure - also known as a pancreaticoduodenectomy - is a complex operation to remove the head of the pancreas, the first part of the small intestine (duodenum), the gallbladder and the bile duct.
  The Whipple procedure is used to treat tumors and other disorders of the pancreas, intestine and bile duct. It is the most often used surgery to treat pancreatic cancer that's confined to the head of the pancreas. After performing the Whipple procedure, your surgeon reconnects the remaining organs to allow you to digest food normally after surgery. Standard of care.
  Major surgery: Additional surgical procedure(s) that is clinically indicated. Standard of care.
Period: Overall Study
Arm/Group | Normal Preoperative Lung Function | Preoperative COPD
Started | 0 | 1
Completed | 0 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Data was not analyzed or disclosed due to subject confidentiality being an issue (n=1). Study terminated due to poor enrollment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Normal Preoperative Lung Function | Preoperative COPD | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Categorical
Sex: Female, Male
Race and Ethnicity Not Collected — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Correlation of AxV-128/Tc Uptake and Fibrinogen
Description: To determine if peri-operative lung injury can be detected with in vivo imaging in patients with COPD
Time Frame: Up to 1 week from initial scan
Population: Study terminated due to poor enrollment. Data was not analyzed or disclosed due to subject confidentiality being an issue (n=1).
Arm/Group | Normal Preoperative Lung Function | Preoperative COPD
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Correlation of AxV-128/Tc Uptake and C-Reactive Protein (CRP)
Description: To determine if peri-operative lung injury can be detected with in vivo imaging in patients with COPD
Time Frame: Up to 1 week from initial scan
Population: as for outcome 1
Arm/Group | Normal Preoperative Lung Function | Preoperative COPD
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Correlation of AxV-128/Tc Uptake and White Blood Cell (WBC) Count
Description: To determine if peri-operative lung injury can be detected with in vivo imaging in patients with COPD
Time Frame: Up to 1 week from initial scan
Population: as for outcome 1
Arm/Group | Normal Preoperative Lung Function | Preoperative COPD
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: AxV-128/Tc Uptake
Description: To determine if peri-operative lung injury can be detected with in vivo imaging in patients with COPD
Time Frame: Up to 1 week from initial scan
Population: as for outcome 1
Arm/Group | Normal Preoperative Lung Function | Preoperative COPD
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Correlation of AxV-128/Tc Uptake and RAGE
Description: To determine if peri-operative lung injury can be detected with in vivo imaging in patients with COPD
Time Frame: Up to 1 week from initial scan
Population: as for outcome 1
Arm/Group | Normal Preoperative Lung Function | Preoperative COPD
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Correlation of AxV-128/Tc Uptake and IL-6
Description: To determine if peri-operative lung injury can be detected with in vivo imaging in patients with COPD
Time Frame: Up to 1 week from initial scan
Population: as for outcome 1
Arm/Group | Normal Preoperative Lung Function | Preoperative COPD
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Correlation of AxV-128/Tc Uptake and Clara-cell 16
Description: To determine if peri-operative lung injury can be detected with in vivo imaging in patients with COPD
Time Frame: Up to 1 week from initial scan
Population: as for outcome 1
Arm/Group | Normal Preoperative Lung Function | Preoperative COPD
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Correlation of AxV-128/Tc Uptake and SP-D
Description: To determine if peri-operative lung injury can be detected with in vivo imaging in patients with COPD
Time Frame: Up to 1 week from initial scan
Population: as for outcome 1
Arm/Group | Normal Preoperative Lung Function | Preoperative COPD
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 1 week from initial scan
Description: Study terminated due to poor enrollment. Data was not analyzed or disclosed due to subject confidentiality being an issue (n=1).
Arm/Group | Normal Preoperative Lung Function | Preoperative COPD
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Study terminated due to poor enrollment. Data was not analyzed or disclosed due to subject confidentiality being an issue (n=1).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-21): https://cdn.clinicaltrials.gov/large-docs/85/NCT02978885/Prot_SAP_000.pdf